CLINICAL TRIAL: NCT01851200
Title: Brentuximab Vedotin (SGN-35) as Salvage Therapy for Males With Advanced and Platinum-resistant Germ-cell Tumors. An Open Label, Single Group, Phase 2 Trial.
Brief Title: Brentuximab Vedotin (SGN-35) as Salvage Treatment for CD30-positive Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Michelangelo (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FM-12-GCT01; 2012-004508-36 (EudraCT Number)
Record Dates: First submitted 2013-04-20; First posted 2013-05-10 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2016-04

CONDITIONS: Germ Cell Cancer
Keywords: Testicular neoplasms; Germ Cell cancers; Embryonal Carcinoma; Metastatic; Brentuximab Vedotin
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms; Carcinoma, Embryonal; Neoplasm Metastasis | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brentuximab Vedotin (Experimental): Intravenous Brentuximab Vedotin at the dose of 1.8 mg/Kg every 3 weeks until disease progression or onset of unacceptable toxicity
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Intravenous Brentuximab Vedotin at the dose of 1.8 mg/Kg every 3 weeks until disease progression or onset of unacceptable toxicity
  Other Names: SGN-35; Adcetris

SUMMARY:
The purpose of the study is to assess the activity of Brentuximab vedotin in refractory germ cell tumors.

DETAILED DESCRIPTION:
Complete responses with third-line or later salvage chemotherapy (CT) for germ cell tumors (GCT) range 0% to 10% and are usually short-lived and nearly all patients (pts) progressing after multiple courses or high-dose CT will ultimately die from progressive disease.

Cluster of Differentiation antigen-30 (CD30) is expressed by untreated embryonal carcinoma (ECA) thus lending support to a rationale for a targeted approach. The investigators retrospectively re-assessed ECA to strongly retain CD30 staining in most cases (>70%), even after multiple courses or high-dose CT. Moreover, a negative prognostic value of CD30 expression by residuals after CT, particularly in the salvage setting, was set. Brentuximab vedotin is an antibody-drug conjugate consisting of the chimeric anti-CD30 antibody chemically conjugated to an antitubulin synthetic analog (MMAE).

Proof of activity will provide rationale for developing first-line chemo-immunotherapy or maintenance immunotherapy for selected high-risk pts. The primary objective of the study will be the activity of Brentuximab vedotin in refractory GCT. Secondary objectives will include safety and survival.

24 pts with biopsy-proven CD30 positive GCT will receive intravenous Brentuximab vedotin at the dose of 1.8 mg/Kg every 3 weeks until disease progression or onset of unacceptable toxicity. Further eligibility requirements will include failure of 2 or 3 platinum-based CT (prior high-dose CT is allowed). All pts will undergo measurement of serum tumor markers, a computed tomography and a positron emission tomography (PET) scan every weeks. An optimal Simon's 2-stage design will be applied. The primary endpoint is the objective response-rate (ORR). An ORR of 5% is not promising, while a 25% rate will be promising. In stage 1, 9 evaluable patients will be accrued. The type I and II error are both set at 10%.

Additional post-treatment tissue will be available for pts undergoing surgery in the treatment time-course. Tissue array blocks will be constructed from samples of all pts. Assessment will include mutational analysis of most-frequently mutated genes. Two serum aliquots will be collected at baseline and during/end of treatment to assess circulating CD30.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years.
* Confirmation of germ cell tumor histology based on pathologic review at the study site.
* Presence of a CD30 positive embryonal carcinoma component.
* Unequivocal progression of measurable disease.
* A minimum of 2 and a maximum of 3 platinum-based chemotherapy lines for metastatic disease EXCEPT for primary mediastinal germ cell tumors where failure of first-line chemotherapy only is accepted.
* Prior high dose chemotherapy with hematopoietic stem cell rescue is allowed.

Exclusion Criteria:

* Failure to meet any of the above inclusion criteria.
* Patients with late-relapse (defined as relapse occurring after at least 2 years from the date of completion of the last chemotherapy regimen) whose disease is completely surgically resectable (and for whom initial surgical extirpation is recommended) are ineligible. Patients with unresectable late disease relapse are eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The number of objective responses (partial and complete responses) according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 integrated with response of serum tumor markers. | Six weeks after the first administration of the study drug.

SECONDARY OUTCOMES:
Progression-Free Survival | 3 months after the initiation of study treatment
Overall Survival | Six months after the initiation of study treatment
Incidence of adverse events related to the study drug | Six weeks after the initiation of the study drug and every 6 weeks thereafter up to 16 weeks.

OTHER OUTCOMES:
Metabolic response to Brentuximab Vedotin measured by means of a Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography (FDG-PET/CT) scan. | Six weeks after the first administration of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro M Gianni, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Roberto Salvioni, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Andrea Necchi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Mi, Italy

REFERENCES:
- See also: Web site of the study Sponsor — http://www.fondazionemichelangelo.org